CLINICAL TRIAL: NCT07114224
Title: Aβ PET and Tau PET Imaging in the Diagnosis and Progression Assessment of Alzheimer's Disease
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: KY20252271
Record Dates: First submitted 2025-08-04; First posted 2025-08-11 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Alzheimer Disease (AD); Cognitive Dysfunction, Cognitive Disorder; PET Imaging
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- normal volunteer group (Experimental)
  Interventions: Diagnostic Test: AV45/AV-1、AV1451 PET
- Alzheimer's disease and cognitive impairment group (Experimental)
  Interventions: Diagnostic Test: AV45/AV-1、AV1451 PET

INTERVENTIONS:
Diagnostic Test: AV45/AV-1、AV1451 PET — Use PET equipment to collect multimodal imaging data. Sixty to ninety minutes after intravenous injection of 3.7 MBq/kg of 18F-AV45 or 18F-AV1, perform PET imaging in list mode to simultaneously collect structural and functional information under the same pathophysiological conditions.
  The next day, perform 18F-AV1451 PET imaging to obtain tau protein distribution information.

SUMMARY:
This prospective study recruited 20 healthy volunteers and 50 patients diagnosed with Alzheimer's disease (AD) and mild cognitive impairment (MCI) according to clinical guidelines. Participants underwent AV45/AV-1 and AV1451 PET imaging to obtain information on Aβ protein deposition, tau protein distribution, and structural and functional information. The study aims to evaluate the value of multimodal imaging features in the diagnosis and progression assessment of AD, providing imaging evidence for novel treatment modalities such as lecanemab therapy and deep cervical vein-lymphatic anastomosis.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-75 years old; Healthy volunteers: males weighing ≥50 kg, females weighing ≥45 kg, with a body mass index (BMI = weight (kg)/height² (m²)) within the range of 19.0-28.0 kg/m² (including boundary values); Cognitive disorders diagnosed clinically according to guidelines include Alzheimer's disease (AD) and mild cognitive impairment (MCI). Diagnostic criteria are as follows: 1) Clinical manifestations include symptoms such as memory impairment, difficulty concentrating, slowed thinking, and poor language skills; 2) Neuropsychological tests show that functions such as memory, attention, thinking, and language are below the normal population level; 3) Blood or cerebrospinal fluid tests show elevated levels of human β-amyloid 1-42, human β-amyloid 1-40, and human phosphorylated tau protein. 4) Exclusion of other factors that may cause cognitive impairment, such as drug or substance abuse, environmental factors, etc.; Signing an informed consent form for PET/MR or PET/CT examinations and voluntarily participating in this study.

Exclusion Criteria:

* Minors, pregnant women, breastfeeding women, individuals with severe liver or kidney dysfunction, and those with a history of allergy to contrast agents or other medications; Diagnosed with viral encephalitis, acute myelitis, idiopathic epilepsy, or antibody-negative AIE; Diagnosed with any major illness; history of alcohol or drug abuse/dependence; History of cardiovascular disease, tumours, blood disorders, or poorly controlled chronic conditions; Contraindications for PET/MR imaging. History of head trauma or surgery; History of other neurological disorders.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-08-15 (Estimated); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
SUVmean | 1 hour from injection of the tracer
  mean of standardized uptake value
VOI | 1 day from injection of the tracer
  volume of interest